CLINICAL TRIAL: NCT05741671
Title: Sonographic Features of Fibroids Before and During Non-surgical Therapy and/or Expectant Management
Acronym: MYOVASC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Marjolein Spiering, Investigator Reseach Office Womens Child Center, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2017.494
Record Dates: First submitted 2023-01-11; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Fibroid Uterus
Keywords: fibroid; power doppler; vascularization
MeSH Terms: conditions — Leiomyoma; Neovascularization, Pathologic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- natural course: To study the value of sonographic features including vascularity in the prediction of fibroids' volume change at follow-up during their (1) natural course or (2) long-term use of exogenous hormone exposure; after initiation of (3) SPRMs or GnRH-analogues treatment or (4) exogenous hormonal exposure; or after (5) embolization or (6) ablation therapy .
  Primary outcome: Natural behaviour - 1 year
  Interventions: Other: Questionnaire
- during long-term use of exogenous hormone exposure: To study the value of sonographic features including vascularity in the prediction of fibroids' volume change at follow-up during their (1) natural course or (2) long-term use of exogenous hormone exposure; after initiation of (3) SPRMs or GnRH-analogues treatment or (4) exogenous hormonal exposure; or after (5) embolization or (6) ablation therapy .
  Primary outcome: Long-term exogenous hormonal exposure - 1 year
  Interventions: Other: Questionnaire
- Selective progesterone receptor modulators treatment or GnRH-analogues treatment: To study the value of sonographic features including vascularity in the prediction of fibroids' volume change at follow-up during their (1) natural course or (2) long-term use of exogenous hormone exposure; after initiation of (3) SPRMs or GnRH-analogues treatment or (4) exogenous hormonal exposure; or after (5) embolization or (6) ablation therapy .
  Primary outcome: SPRMs or GnRH-analogues - 3 months
  Interventions: Other: Questionnaire
- after initiation exogenous hormonal exposure: To study the value of sonographic features including vascularity in the prediction of fibroids' volume change at follow-up during their (1) natural course or (2) long-term use of exogenous hormone exposure; after initiation of (3) SPRMs or GnRH-analogues treatment or (4) exogenous hormonal exposure; or after (5) embolization or (6) ablation therapy .
  Primary outcome: Initiation of exogenous hormonal exposure - 1 year
  Interventions: Other: Questionnaire
- embolization therapy: To study the value of sonographic features including vascularity in the prediction of fibroids' volume change at follow-up during their (1) natural course or (2) long-term use of exogenous hormone exposure; after initiation of (3) SPRMs or GnRH-analogues treatment or (4) exogenous hormonal exposure; or after (5) embolization or (6) ablation therapy .
  Primary outcome: Embolization - 6 months
  Interventions: Other: Questionnaire
- ablation therapy: To study the value of sonographic features including vascularity in the prediction of fibroids' volume change at follow-up during their (1) natural course or (2) long-term use of exogenous hormone exposure; after initiation of (3) SPRMs or GnRH-analogues treatment or (4) exogenous hormonal exposure; or after (5) embolization or (6) ablation therapy .
  Primary outcome: Ablation therapy - 6 months
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Extra in the context of the study are questionnaires which last a maximum of 5-15 minutes. The treatment considering the fibroid(s) is independent of this research. the Also the outcome measures include vaginal ultrasound, questionaires and a hemoglobin test. These measurements are applied in daily practice, as standard care.

SUMMARY:
Rationale: 20-30% of women of reproductive age have leiomyomas, causing symptoms like dysmenorrhea and pelvic pain which both effect quality of life.[1-4] The natural behaviour of uterine fibroids is to grow between 7 to 84% in 3 to 12 months.[5-7] Non-surgical options to treat uterine fibroids are non-hormonal or hormonal medical therapies and minimally invasive interventional radiologic techniques. Exogenous hormone exposure including COC, POP or Mirena give in conflicting literature minimal growth to 60% volume shrinkage. [8, 9]] Selective progesterone receptor modulators (SPRM) eg. Esmya and GnRH-analogues intent to reduce fibroids volume after several months; GnRH-agonists provide a 31-63% shrinkage and less frequently applied GnRH-antagonists 14.3 - 42.7%.[10-16] Esmya gives a volume reduction varying between 10 to 48%.[17] Radiological technique like embolization decreases dominant fibroid volume with 40-70%.[1, 18-22] UAE fails in case of devascularized or minimal vascularized fibroids.[23] Ablation techniques show shrinkage up to a maximum of 90% depending e.g. which treatment.[24-41] Clear prognostic models to predict the effect on fibroid related symptoms and volume reduction are lacking. We postulate higher vascularity to be related to 1) larger fibroid growth during the natural course or during exogenous hormonal exposure; 2) more effective shrinkage during progestogens, GnRH-analogues, SPRM and UAE; but 3) less effective after ablation therapy.

Objectives: To study the value of sonographic features including vascularity in the prediction of fibroids' volume change at follow-up during their (1) natural course or (2) long-term use of exogenous hormone exposure; after initiation of (3) SPRM or GnRH-analogues treatment or (4) exogenous hormonal exposure; or after (5) embolization or (6) ablation therapy.

Study design: Observational cohort study during 5 years in the outpatient clinic.

Patientselection: Women ≥18 years with 1 to 3 fibroids with a maximal diameter ≥ 3cm and ≤ 10cm diagnosed on ultrasound examination, planned for expectant or non-surgical management. Study objectives: The primary outcome is volume reduction after 3 to 12 month depending on the study group. The secondary outcome include UFS-QOL, EQ-5D score, PBAC, hemoglobin level, treatment failure rate and (re)intervention rate.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: No risks are associated with the participation of this observational study since the outcome measures include vaginal ultrasound, questionaires and a hemoglobin test. These measurements are also applied in daily practice, the burden for the patient is time. Extra in the context of the study are questionnaires which last a maximum of 5-15 minutes. The treatment considering the fibroid(s) is independent of this research.

ELIGIBILITY:
Inclusion Criteria:

* 1 to 3 fibroids
* maximal diameter ≥1.5 cm and ≤ 10 cm
* diagnosed on ultrasound examination with informed consent
* planned for expectant management or non-surgical management in the follwing groups:

  1. Women with uterine fibroids without treatment (during natural course);
  2. Women with uterine fibroids using exogenous hormone exposure for at least 3 months: e.g. COC, POP, DP or LNG-IUD;
  3. Women with uterine fibroids before and after/during treatment with SPRMs or GnRH-analogues;
  4. Women with uterine fibroids before and after/during treatment with exogenous hormones;
  5. Women with uterine fibroids before and after embolization;
  6. Women with uterine fibroids before and after ablation therapy*.

     * In case of embolization or ablation: inclusion in case of multiple fibroids is allowed, if ≥ 1 fibroid is accessible for transvaginal ultrasound.

Exclusion Criteria:

* Any fibroid treatment in the last 3 months in case of (3) SPRMs or GnRH-analogues (except for exogenous hormone exposure) or (1) no treatment Age < 18 years
* Fibroids not accessible for transvaginal ultrasonography
* Suspicion for malignancy
* Postmenopausal
* Severe adenomyosis
* Pregnancy
* Contra-indication for the planned treatment
* Use of aromatase inhibitors or tamoxifen Infertility treatment with use of clomifene and/or follicle-stimulating hormone Breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Fibroids are uterine-related
Study Population: Women pre- to perimenopausal with uterus myomatosis. Uterus myomatosis occurs in 20-30% of women of reproductive age.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Volume change | Baseline, 3 and 12 months, in embolization and ablation group after 6 months
  Three directions on 2D ultrasound in centimeters.

SECONDARY OUTCOMES:
Questionnaire Utreine Fibroid Specific Quality of Life | Baseline, 3, 12 and 24 months, in embolization and ablation group after 6 months
  UFS-Qol. Total health-related quality of life (29 items, 29-145 points). Or seven subscales: 'symptom severity' (8 items, 8-40 points), 'concern' (5 items, 5-25 points), 'activities' (7 items, 7-35 points), 'energy/mood' (7 items, 7-35 points), 'control' (5 items, 5-25 points), 'self-conscious' (3 items, 3-15 points), 'sexual function' (2 items, 2-10 points). The higher, the lower the quality of life.
Questionnaire EuroQol 5 Dimensions | Baseline, 3, 12 and 24 months, in embolization and ablation group after 6 months
  EQ-5D. Range 0 - 1. The higher, the lower the quality of life.
Questionnaires Picterial Bloodloss Assessment Chart | Baseline, 3, 12 and 24 months, in embolization and ablation group after 6 months
  PBAC. Range 0 to no maximum. PBAC > 150 is heavy menstrual bleeding. The higher, the more bloodloss.
Questionnaire re-intervention rate | Baseline, 3, 12 and 24 months, in embolization and ablation group after 6 months
  Percentage of patients who underwent re-intervention (e.g. embolization, operation, etc) for their fibroid(s) in follow-up period. Range: 0-100%, the higher, the more re-interventions.
Questionnaire treatment failure rate | Baseline, 3, 12 and 24 months, in embolization and ablation group after 6 months
  Percentage of patients who started additional treatment (e.g. medication, etc) for their fibroid(s) in follow-up period. Range: 0-100%, the higher, the more treatment failures.
Haemoglobin | Baseline, 3 and 12 months, in embolization and ablation group after 6 months
  According to local protocol, standard care, mmol/L (range 0-20). A lower haemoglobin level corresponds with more menstrual bloodloss and/or anemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No